CLINICAL TRIAL: NCT05651594
Title: A Phase 2 Trial of Chemotherapy, Pembrolizumab, and Propranolol in Advanced Esophageal/Gastroesophageal Junction Adenocarcinoma Patients
Brief Title: Propranolol in Combination With Pembrolizumab and Standard Chemotherapy for the Treatment of Unresectable Locally Advanced or Metastatic Esophageal or Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 2734222; NCI-2022-09209 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 2734222 (Other: Roswell Park Cancer Institute); W81XWH2210916 (Other Grant/Funding Number: DOD)
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Clinical Stage II Esophageal Adenocarcinoma AJCC v8; Clinical Stage III Esophageal Adenocarcinoma AJCC v8; Clinical Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IV Esophageal Adenocarcinoma AJCC v8; Clinical Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Locally Advanced Esophageal Adenocarcinoma; Locally Advanced Gastroesophageal Junction Adenocarcinoma; Metastatic Esophageal Adenocarcinoma; Metastatic Gastroesophageal Junction Adenocarcinoma; Unresectable Esophageal Adenocarcinoma; Unresectable Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — Biopsy; Specimen Handling; Fluorouracil; dehydroftorafur; Leucovorin; Oxaliplatin; pembrolizumab; Propranolol; propranolol CR

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (mFOLFOX6, pembrolizumab, propranolol) (Experimental): Patients receive mFOLFOX6 (leucovorin IV, oxaliplatin IV, and fluorouracil IV), pembrolizumab IV, and propranolol PO on study. Patients also undergo tumor biopsy during screening and CT scans and collection of blood samples during screening and on study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin; Biological: Pembrolizumab; Drug: Propranolol Hydrochloride; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biopsy — Undergo tissue collection
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scans
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Leucovorin — Given IV
  Other Names: Folinic acid
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Propranolol Hydrochloride — Given PO
  Other Names: Inderal; Innopran XL
Other: Questionnaire Administration — Perceived Stress Scale

SUMMARY:
This phase II trial tests what effects the addition of propranolol to pembrolizumab and standard chemotherapy (mFOLFOX) may have on response to treatment in patients with esophageal or gastroesophageal junction cancer that cannot be removed by surgery and has spread to nearby tissue or lymph nodes (unresectable locally advanced) or has spread from where it first started (primary site) to other places in the body (metastatic). Propranolol is a drug that is classified as a beta-blocker. Beta-blockers affect the heart and circulation (blood flow through arteries and veins). Cancer patients may be under a tremendous amount of stress with elevated levels of norepinephrine (a hormone produced by the adrenal glands in response to stress). Increased adrenergic stress may dampen the immune system, which beta-blockers, like propranolol, may be able to counteract. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in the standard chemotherapy regimen, mFOLFOX (leucovorin, fluorouracil and oxaliplatin) work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Adding propranolol to pembrolizumab and standard mFOLFOX chemotherapy may increase the effectiveness of the pembrolizumab + mFOLFOX regimen.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the clinical efficacy of propranolol in combination with pembrolizumab and standard chemotherapy in frontline metastatic esophageal or gastroesophageal junction (GEJ) adenocarcinoma.

SECONDARY OBJECTIVE:

I. To evaluate the progression-free survival, overall survival, overall response rate, and safety profile of the combination of pembrolizumab and propranolol with standard chemotherapy.

EXPLORATORY OBJECTIVE:

I. To correlate baseline or changes in the levels of biomarkers (e.g., like, peripheral T-cell subsets/myeloid-derived suppressor cells [MDSC]/cytokines), perceived stress and exercise Perceived Stress Scale (PSS) with efficacy (overall response rate [ORR], progression-free survival [PFS], overall survival [OS]), and chronotropic effect of exercise.

OUTLINE:

Patients receive mFOLFOX6 (leucovorin intravenously [IV], oxaliplatin IV, and fluorouracil IV), pembrolizumab IV, and propranolol orally (PO) on study. Patients also undergo tumor biopsy during screening and computed tomography (CT) scans and collection of blood samples during screening and on study.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years of age.
* Participants must be newly diagnosed, treatment-naive with unresectable locally advanced or metastatic esophageal/gastroesophageal junction (GEJ) adenocarcinoma. Any prior systemic treatment for resectable disease must be six months or before. Prior PD-1/PD-L1 treatment is allowed as long as the treatment was completed more than 1 year ago.
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Available archival Formalin-Fixed Paraffin-Embedded (FFPE) from a prior biopsy collected within 1 year or, participant must be willing to have a tissue biopsy taken prior to start of study treatment.
* Have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria present.
* Platelet >= 75,000/uL
* Hemoglobin >= 8 g/dL (without transfusion in the past 14 days)
* Absolute Neutrophil Count (ANC) >= 1500/uL
* Creatinine clearance (Cockcroft Gault) >= 30 mL/min
* Total bilirubin: =< 2 × upper limit of normal (ULN) OR direct bilirubin =< ULN for participants with total bilirubin levels > 2 × ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase) (SGOT) and alanine transaminase (ALT) (serum glutamic-pyruvic transaminase) (SGPT) =< 3 X institutional ULN (=< 5 × ULN for participants with liver metastases)
* Participants of child-bearing potential must have a negative pregnancy test at study entry and then agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability to swallow and retain oral medication. If a patient is not able to swallow or is experiencing dysphagia that limits ability to swallow oral medication, they are still eligible for study provided they can swallow liquid formula propranolol or have an enteric feeding tube placed which will permit administration of crushed tablets or liquid formula propranolol. Liquid and tablet formulations may be used interchangeably for patients in the event of a shortage of either formulation
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* Patients with HER 2-positive cancer.
* Patients with active, untreated central nervous system metastases or leptomeningeal disease.
* Patients with active autoimmune disease, requiring ongoing immunosuppressive therapy or history of transplantation.

  * Patients currently treated with systemic immunosuppressive agents: If a patient is currently on steroids, they must be on a steroid dose less than or equal to an equivalent prednisone dose of 10 mg daily.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required treatment.
* Has a concurrent Human Immunodeficiency Virus (HIV) infection.
* Concurrent active Hepatitis B (defined as Hepatitis B virus surface antigen [HBsAg] positive and/or detectable Hepatitis B virus [HBV] deoxyribonucleic acid DNA) and Hepatitis C virus (defined as anti-HCV antibody [Ab] positive and detectable HCV ribonucleic acid [RNA]) infection. Note: Hepatitis B and C screening tests are not required unless known history of HBV and HCV infection.
* Participants that are already on beta-adrenergic (B-AR) blockers for various indications.
* Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (=<2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or nursing female participants, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.
* Other active cancers that require systemic treatment.
* Contraindications to the use of beta-blockers, e.g.: uncontrolled depression, unstable angina pectoris, uncontrolled heart failure ( Grade III or IV), hypotension (systolic blood pressure <100 mmHg), severe asthma or chronic obstructive pulmonary disease (COPD), uncontrolled type I or type II diabetes mellitus (HbA1C > 8.5 or fasting plasma glucose > 160 mg/dl at screening), symptomatic peripheral arterial disease or Raynaud's syndrome, untreated pheochromocytoma etc.
* Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of trial treatment and while participating in the trial. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster etc.
* Unwilling or unable to follow protocol requirements.
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Within 6 months of initiating combination therapy
  Efficacy of pembrolizumab in combination with propranolol with standard chemotherapy measured by ORR by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, which is treated as a dichotomous variable and will be summarized using frequencies and relative frequencies.

SECONDARY OUTCOMES:
Incidence of toxicities and adverse events | Up to 30 days after the last intervention
  Will be assessed as per Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.
Progression-free survival | Initiation of the study treatment regimen to disease progression or death from any cause, assessed up to 2 years
  Will be summarized using standard Kaplan Meier methods.
Overall survival | Treatment initiation until death from any cause, assessed up to 2 years
  Will be summarized using standard Kaplan Meier methods.
ORR | Within 6 months of initiating combination therapy
  ORR as determined by Immune-Modified (i)RECIST.

CONTACTS AND LOCATIONS:
Overall Officials: Kannan Thanikachalam, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States